CLINICAL TRIAL: NCT00553501
Title: A Phase II Trial of Extended Induction Epratuzumab (Anti-CD22 Monoclonal Antibody) (CALGB IND #XXXXX) Plus Rituximab in Previously Untreated Follicular Non-Hodgkin's Lymphoma (NHL)
Brief Title: Epratuzumab and Rituximab in Treating Patients With Previously Untreated Follicular Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-50701; U10CA031946 (NIH); CALGB-50701; CDR0000572604 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Results first posted 2014-07-24 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lymphoma
Keywords: stage II grade 1 follicular lymphoma; stage II grade 2 follicular lymphoma; stage II grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — epratuzumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Epratuzumab Plus Rituximab (Experimental): Induction Therapy (Month 1): Epratuzumab 360 mg/m^2 by IV days 1, 8, 15 & 22; Rituximab 375 mg/m^2 by IV day 3, 8, 15 & 22
  Extended Induction (Weeks 12, 20, 28 & 36) Epratuzumab 360 mg/m^2 by IV weeks 12, 20, 28 & 36; Rituximab 375 mg/m^2 by IV weeks 12, 20, 28 & 36
  Interventions: Biological: epratuzumab; Biological: rituximab

INTERVENTIONS:
Biological: epratuzumab — Days 1, 8, 15, 22 and weeks 12, 20, 28, & 36: 360mg/sq m IV
Biological: rituximab — Day 3, 8, 15, 22 and weeks 12, 20, 28, & 36: 375mg/sq m IV

SUMMARY:
RATIONALE: Monoclonal antibodies, such as epratuzumab and rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving epratuzumab and rituximab together may be more effective in treating follicular non-Hodgkin lymphoma.

PURPOSE: This phase II trial is studying how well giving epratuzumab together with rituximab works in treating patients with previously untreated follicular non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate (overall and complete) after extended induction therapy comprising epratuzumab and rituximab in patients with previously untreated CD20+ follicular non-Hodgkin lymphoma (NHL).
* To determine the time to progression after extended induction therapy comprising epratuzumab and rituximab in patients with previously untreated CD20+ follicular NHL.

Secondary

* To determine the toxicity profile of epratuzumab and rituximab in patients with previously untreated CD20+ follicular NHL.
* To establish whether the therapeutic effects of the combination of epratuzumab and rituximab are sufficiently promising to warrant evaluation in a subsequent randomized trial (in comparison to rituximab alone).
* To determine the relationship between the change in fludeoxyglucose F 18 uptake early after epratuzumab and rituximab treatment with response rate and time to progression.

OUTLINE:

* Induction therapy (month 1): Patients receive epratuzumab IV over 5-30 minutes on days 1, 8, 15, and 22 and rituximab IV on days 3, 8, 15, and 22 in the absence of disease progression or unacceptable toxicity.
* Extended induction therapy (months 3, 5, 7, and 9): Patients receive epratuzumab IV over 5-30 minutes followed by rituximab IV in weeks 12, 20, 28, and 36 in the absence of disease progression or unacceptable toxicity.

Patients receive fludeoxyglucose F 18 (FDG) subcutaneously and undergo positron emission tomography at baseline and after induction therapy to assess the degree of FDG uptake.

After completion of study treatment, patients are followed every 4 months for 2 years then every 6 months for up to 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically* confirmed follicular non-Hodgkin lymphoma (NHL)

  * Previously untreated disease
  * WHO classification grade 1, 2, or 3a (> 15 centroblasts per high power field with centrocytes present) that is stage III, IV, or bulky (i.e., single mass ≥ 7 cm in any unidimensional measurement) stage II disease NOTE: *Bone marrow biopsies as the sole means of diagnosis are not acceptable, but they may be submitted in conjunction with nodal biopsies; fine-needle aspirates are not acceptable for diagnosis
* Confirmed CD20 antigen expression by flow cytometry or immunohistochemistry
* Measurable disease by physical examination or imaging studies

  * Any tumor mass > 1 cm is acceptable
  * No nonmeasurable disease only, including any of the following:

    * Bone lesions
    * Ascites
    * Pleural/pericardial effusion
    * Lymphangitis cutis/pulmonis
    * Bone marrow (involvement by NHL should be noted)
* No known CNS involvement by lymphoma
* Required to participate in companion FDG-PET imaging study CALGB 580701

PATIENT CHARACTERISTICS:

* ECOG performance status ≤ 2
* Absolute neutrophil count ≥ 1,000/μL
* Platelet count ≥ 50,000/μL
* Patients with HIV infection are eligible provided they meet the following criteria:

  * No evidence of coinfection with hepatitis B or C
  * CD4+ cell count ≥ 400/mm^3
  * No evidence of resistant strains of HIV
  * If not on anti-HIV therapy, HIV viral load < 10,000 copies HIV RNA/mL
  * If on anti-HIV therapy, HIV viral load < 50 copies HIV RNA/mL
  * No history of AIDS-defining conditions
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after completion of study therapy
* No known Human Anti-Chimeric Antibody (HACA)-positivity

PRIOR CONCURRENT THERAPY:

* No prior therapy for NHL including chemotherapy, radiotherapy, or immunotherapy (e.g., monoclonal antibody-based therapy)
* More than 2 weeks since prior corticosteroids except for maintenance therapy for non-malignant disease
* No concurrent dexamethasone or other steroids as antiemetics except for the following circumstances:

  * Treatment of acute infusion reactions according to institutional procedures
* No concurrent hormonal therapy except steroids for adrenal failure OR hormones for non-disease-related conditions (e.g., insulin for diabetes)
* No other concurrent chemotherapeutic agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Grant, MD, Study Chair — University of Vermont
Locations (43):
- United States (43):
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Union Hospital Cancer Program at Union Hospital, Elkton MD, Maryland
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Danville Regional Medical Center, Danville, Virginia
  - Ravenel Oncology Center at Memorial Hospital of Martinsville and Henry County, Martinsville, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia

REFERENCES:
- [Result] Grant BW, Jung SH, Johnson JL, Kostakoglu L, Hsi E, Byrd JC, Jones J, Leonard JP, Martin SE, Cheson BD. A phase 2 trial of extended induction epratuzumab and rituximab for previously untreated follicular lymphoma: CALGB 50701. Cancer. 2013 Nov 1;119(21):3797-804. doi: 10.1002/cncr.28299. Epub 2013 Aug 6. PMID 23922187
- [Derived] Rutherford SC, Yin J, Pederson L, Perez Burbano G, LaPlant B, Shadman M, Li H, LeBlanc ML, Kenkre VP, Hong F, Blum KA, Dockter T, Martin P, Jung SH, Grant B, Rosenbaum C, Ujjani C, Barr PM, Unger JM, Cheson BD, Bartlett NL, Kahl B, Friedberg JW, Mandrekar SJ, Leonard JP. Relevance of Bone Marrow Biopsies for Response Assessment in US National Cancer Institute National Clinical Trials Network Follicular Lymphoma Clinical Trials. J Clin Oncol. 2023 Jan 10;41(2):336-342. doi: 10.1200/JCO.21.02301. Epub 2022 Jul 5. PMID 35787017
- [Derived] Lansigan F, Barak I, Pitcher B, Jung SH, Cheson BD, Czuczman M, Martin P, Hsi E, Schoder H, Smith S, Bartlett NL, Leonard JP, Blum KA. The prognostic significance of PFS24 in follicular lymphoma following firstline immunotherapy: A combined analysis of 3 CALGB trials. Cancer Med. 2019 Jan;8(1):165-173. doi: 10.1002/cam4.1918. Epub 2018 Dec 21. PMID 30575311

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2008 and July 2009, 60 participants were recruited.
Pre-assignment Details: One participant was deemed ineligible and excluded from all analyses per study design.
Period: Overall Study
Arm/Group | Epratuzumab Plus Rituximab
Started | 59
Completed | 55
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Epratuzumab Plus Rituximab
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 54 [32 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 54
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Overall Response
Description: Overall response is defined as achievement of a complete response (CR) or partial response (PR) as defined by the Revised Response Criteria for Malignant Lymphoma.
  CR: complete disappearance of all detectable disease PR: >=50% decrease in the sum of the product of diameters of indicator lesions
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Epratuzumab Plus Rituximab
Number analyzed (Participants) | 59
participants
  Complete Response | 25
  Partial Response | 27

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) was defined as the time from registration to progression or death of any cause. Progression free and alive patients were censored at the date of last follow-up. The median PFS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 10 years)
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Epratuzumab Plus Rituximab
Number analyzed (Participants) | 59
years | 3.5 [2.6 to 4.4]

3. Post Hoc Outcome: 3-Year Overall Survival
Description: Percentage of participants who were alive at 3 years. The 3 year survival, with 95% confidence interval, was estimated using the Kaplan Meier method.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Epratuzumab Plus Rituximab
Number analyzed (Participants) | 59
percentage of participants | 91 [80 to 96]

ADVERSE EVENTS:
Arm/Group | Epratuzumab Plus Rituximab
Serious Adverse Events (participants affected / at risk) | 10/59
Other Adverse Events (participants affected / at risk) | 58/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epratuzumab Plus Rituximab (N=59)
Hemoglobin decreased (Blood and lymphatic system disorders) | 6 (7)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 3 (4)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 8 (9)
Fever (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Visceral edema (General disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Peripheral nerve infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 2 (2)
Cardiac troponin I increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 2 (2)
Laboratory test abnormal (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 5 (6)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 2 (3)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Mini mental status examination abnormal (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epratuzumab Plus Rituximab (N=59)
Hemoglobin decreased (Blood and lymphatic system disorders) | 15 (37)
Lymph node pain (Blood and lymphatic system disorders) | 7 (13)
Cardiac disorder (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 1 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (3)
Eye disorder (Eye disorders) | 1 (2)
Vision blurred (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 10 (14)
Constipation (Gastrointestinal disorders) | 11 (21)
Diarrhea (Gastrointestinal disorders) | 5 (10)
Dry mouth (Gastrointestinal disorders) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (3)
Gingival pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 21 (29)
Stomach pain (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 6 (8)
Chills (General disorders) | 8 (8)
Edema limbs (General disorders) | 6 (10)
Fatigue (General disorders) | 35 (100)
Fever (General disorders) | 11 (15)
Flu-like symptoms (General disorders) | 1 (1)
General symptom (General disorders) | 1 (1)
Pain (General disorders) | 6 (9)
Cytokine release syndrome (Immune system disorders) | 5 (9)
Hypersensitivity (Immune system disorders) | 2 (4)
Immune system disorder (Immune system disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 6 (11)
Urinary tract infection (Infections and infestations) | 3 (3)
Vaginal infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 7 (19)
Alkaline phosphatase increased (Investigations) | 4 (12)
Aspartate aminotransferase increased (Investigations) | 11 (22)
Blood bilirubin increased (Investigations) | 13 (29)
Creatinine increased (Investigations) | 4 (15)
Laboratory test abnormal (Investigations) | 5 (12)
Leukocyte count decreased (Investigations) | 12 (28)
Lymphocyte count decreased (Investigations) | 10 (18)
Neutrophil count decreased (Investigations) | 6 (13)
Platelet count decreased (Investigations) | 12 (24)
Weight loss (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Blood glucose increased (Metabolism and nutrition disorders) | 22 (60)
Blood uric acid increased (Metabolism and nutrition disorders) | 4 (6)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (11)
Serum calcium decreased (Metabolism and nutrition disorders) | 7 (13)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 7 (11)
Serum phosphate decreased (Metabolism and nutrition disorders) | 5 (12)
Serum potassium decreased (Metabolism and nutrition disorders) | 9 (11)
Serum potassium increased (Metabolism and nutrition disorders) | 9 (14)
Serum sodium decreased (Metabolism and nutrition disorders) | 13 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (16)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 5 (6)
Dysgeusia (Nervous system disorders) | 2 (3)
Extrapyramidal disorder (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (13)
Memory impairment (Nervous system disorders) | 1 (2)
Neuralgia (Nervous system disorders) | 1 (5)
Neurological disorder NOS (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (11)
Tremor (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (8)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 8 (17)
Libido decreased (Psychiatric disorders) | 1 (2)
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (2)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 4 (4)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (11)
Rash desquamating (Skin and subcutaneous tissue disorders) | 6 (7)
Skin disorder (Skin and subcutaneous tissue disorders) | 5 (6)
Sweating (Skin and subcutaneous tissue disorders) | 5 (8)
Flushing (Vascular disorders) | 2 (3)
Hot flashes (Vascular disorders) | 5 (10)
Hypertension (Vascular disorders) | 4 (8)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less